CLINICAL TRIAL: NCT06566599
Title: A Retrospective Review of the Utilization of Preimplantation Genetic Testing for Aneuploidy (PGT-A) in Couples With Non-obstructive Azoospermia (NOA)
Brief Title: Preimplantation Genetic Testing for Aneuploidy (PGT-A) in Couples With Non-obstructive Azoospermia (NOA)
Status: Enrolling by invitation | Type: Observational
Sponsor: Inception Fertility Research Institute, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: INC-IIS-2024-005
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Non-obstructive Azoospermia; Male Infertility
Keywords: IVF; PGT-A; TESE; PESE
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Objective: To examine the rate of embryo aneuploidy in patients with non-obstructive azoospermia (NOA) who utilize in-vitro fertilization (IVF)/intracytoplasmic sperm injection (ICSI) and compare live birth rates with the utilization of preimplantation genetic testing for aneuploidy (PGT-A) vs non PGT-A.

DETAILED DESCRIPTION:
Preimplantation genetic testing for aneuploidy (PGT-A) facilitates selection of euploid embryos for transfer and may improve outcomes in select couples when the female partner is 35 or older. While embryonic aneuploidy is known to be associated with maternal risk factors such as advanced age, the male factors contributing to aneuploidy are not as clear. Severe male factor infertility is associated with various genetic causes, including karyotypic abnormalities. One retrospective analysis of 668 infertile patients diagnosed with various nonobstructive spermatogenic defects using high resolution Giemsa banding chromosome analysis and/or fluorescence in situ hybridization revealed constitutional chromosomal abnormalities in 55 (8.2%) patients. The observed incidence was almost 20-fold greater than what is reported in healthy fertile men (0.37%). This study correlated cytogenetic aberrations with male reproductive phenotypes and noted that sex chromosome aneuploidy was the most common finding in azoospermia (AS) cases, accounting for about 9%, with Klinefelter syndrome (47, XXY karyotype and variants) accounting for 4% of all infertile males. Notably, the 47, XXY karyotype was detected at a considerably higher rate in men with AS vs oligospermia (OS) (27 of 668 or 9.1% vs 3 of 365 or 0.8%). Little is known about the impact of constitutional aneuploidy on embryonic aneuploidy rates after fertilization with surgically extracted sperm. Another study examined the impact of severe male factor infertility in 326 cycles on aneuploidy in embryos and found significant increases in embryo aneuploidy and higher mosaicism rates in cases using testicular sperm from patients with severe male factor infertility as compared to non-male factor controls. This study found that the statistically significant affected chromosomes were 2, 10, 11, 17, 21 and sex chromosomes. While sperm chromosomal aneuploidy are consistently higher in severe male factor infertility, the impact on IVF outcomes and potential benefits of PGT-A are unclear. Additionally, data on differences in aneuploidy rates between OA and NOA are mixed. Further research is warranted to help facilitate appropriate counseling of affected couples and better understand the role of PGT-A in severe male-factor infertility treatment. We will conduct a retrospective chart review to examine the rates of aneuploidy in embryos resulting from ICSI with surgically extracted sperm in patients with NOA and OA and characterize the chromosomes commonly affected in identified aneuploid embryos.

ELIGIBILITY:
Inclusion Criteria:

* Couples who have undergone in vitro fertilization (IVF) with intracytoplasmic sperm injection (ICSI) with or without pre-implantation genetic testing for aneuploidy (PGT-A) at a fertility clinic in The Prelude Network (US sites only).
* Male partner has diagnosis of non-obstructive azoospermia or obstructive azoospermia.
* Male partner has undergone surgical sperm extraction.

Exclusion Criteria:

* not applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Couples who have undergone IVF/ICSI with or without pre-implantation genetic testing for aneuploidy (PGT-A) at a fertility clinic in The Prelude Network (US sites only).
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Aneuploidy rate | 1 year
  Frequency of aneuploidy result in embryos
Chromosomes associated with aneuploidy | 1 year
  Compare types of embryonic aneuploidy in male factor patients to advanced maternal age patients

SECONDARY OUTCOMES:
Live birth rate | 1 year
  The frequency of live birth following embryo transfer.
Clinical pregnancy rate | 1 year
  The frequency of intrauterine pregnancy (IUP) as confirmed by ultrasound post embryo transfer.
Fertilization rate | 1 year
  The calculated rate of successful fertilization of egg, defined as presence of 2 pronuclei (2PN) on day 1 check post fertilization, to number of eggs where fertilization was attempted.

CONTACTS AND LOCATIONS:
Locations (1):
- Inception Fertility Research Institute, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be available to other researchers.

REFERENCES:
- [Background] Munne S, Kaplan B, Frattarelli JL, Child T, Nakhuda G, Shamma FN, Silverberg K, Kalista T, Handyside AH, Katz-Jaffe M, Wells D, Gordon T, Stock-Myer S, Willman S; STAR Study Group. Preimplantation genetic testing for aneuploidy versus morphology as selection criteria for single frozen-thawed embryo transfer in good-prognosis patients: a multicenter randomized clinical trial. Fertil Steril. 2019 Dec;112(6):1071-1079.e7. doi: 10.1016/j.fertnstert.2019.07.1346. Epub 2019 Sep 21. PMID 31551155
- [Background] Yatsenko AN, Yatsenko SA, Weedin JW, Lawrence AE, Patel A, Peacock S, Matzuk MM, Lamb DJ, Cheung SW, Lipshultz LI. Comprehensive 5-year study of cytogenetic aberrations in 668 infertile men. J Urol. 2010 Apr;183(4):1636-42. doi: 10.1016/j.juro.2009.12.004. Epub 2010 Feb 20. PMID 20172548
- [Background] Ravel C, Berthaut I, Bresson JL, Siffroi JP; Genetics Commission of the French Federation of CECOS. Prevalence of chromosomal abnormalities in phenotypically normal and fertile adult males: large-scale survey of over 10,000 sperm donor karyotypes. Hum Reprod. 2006 Jun;21(6):1484-9. doi: 10.1093/humrep/del024. Epub 2006 Feb 16. PMID 16484311
- [Background] Calogero AE, Burrello N, De Palma A, Barone N, D'Agata R, Vicari E. Sperm aneuploidy in infertile men. Reprod Biomed Online. 2003 Apr-May;6(3):310-7. doi: 10.1016/s1472-6483(10)61850-0. PMID 12735865
- [Background] Rodrigo L, Meseguer M, Mateu E, Mercader A, Peinado V, Bori L, Campos-Galindo I, Milan M, Garcia-Herrero S, Simon C, Rubio C. Sperm chromosomal abnormalities and their contribution to human embryo aneuploidy. Biol Reprod. 2019 Dec 24;101(6):1091-1101. doi: 10.1093/biolre/ioz125. PMID 31318411
- [Background] Asoglu MR, Celik C, Serefoglu EC, Findikli N, Bahceci M. Preimplantation genetic testing for aneuploidy in severe male factor infertility. Reprod Biomed Online. 2020 Oct;41(4):595-603. doi: 10.1016/j.rbmo.2020.06.015. Epub 2020 Jun 27. PMID 32763130
- [Background] Platteau P, Staessen C, Michiels A, Tournaye H, Van Steirteghem A, Liebaers I, Devroey P. Comparison of the aneuploidy frequency in embryos derived from testicular sperm extraction in obstructive and non-obstructive azoospermic men. Hum Reprod. 2004 Jul;19(7):1570-4. doi: 10.1093/humrep/deh306. Epub 2004 May 13. PMID 15142999
- [Background] Kahraman S, Sahin Y, Yelke H, Kumtepe Y, Tufekci MA, Yapan CC, Yesil M, Cetinkaya M. High rates of aneuploidy, mosaicism and abnormal morphokinetic development in cases with low sperm concentration. J Assist Reprod Genet. 2020 Mar;37(3):629-640. doi: 10.1007/s10815-019-01673-w. Epub 2020 Jan 4. PMID 31901112